CLINICAL TRIAL: NCT05450900
Title: Can Biotin Supplementation be Used to Mask hCG Abuse?
Acronym: hCG
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sports Medicine Research and Testing Laboratory (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SMRTL-2022_01
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — Chorionic Gonadotropin; Ovidrel; Biotin; Capsules

STUDY DESIGN:
Intervention Model Description: One cohort receives active drug ovidrel plus biotin supplementation One cohort receives active drug ovidrel plus a placebo
Who Masked: Participant
Masking Description: Every other enrollee
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Active Comparator): hCG plus biotin supplement
  Interventions: Drug: Choriogonadotropin Alpha; Dietary Supplement: biotin
- Cohort 2 (Placebo Comparator): hCG plus placebo supplement
  Interventions: Drug: Choriogonadotropin Alpha; Other: Microcellulose filler

INTERVENTIONS:
Drug: Choriogonadotropin Alpha — drug, active
  Other Names: ovidrel; hCG
Dietary Supplement: biotin — supplement, oral
  Other Names: vitamin B7
  Arms: Cohort 1
Other: Microcellulose filler — supplement, oral
  Other Names: placebo, capsules
  Arms: Cohort 2

SUMMARY:
This sponsor is an anti-doping laboratory tasked with testing athlete samples for prohibited substances by the World Anti-Doping Agency and other agencies.

This study is intended to measure:

1. Urinary/serum hCG (human chorionic gonadotropin) and urinary biotin concentrations in both treatment groups before, during, and after hCG intervention using standard immunoassay methods
2. To monitor hCG in both treatment groups before and after diafiltration of urine samples prior to analysis
3. To compare urinary and serum detectability (detection window, sensitivity) of hCG abuse in the hCG-only group compared to the hCG + biotin group

DETAILED DESCRIPTION:
hCG, or human chorionic gonadotropin, is a protein hormone primarily produced in females by trophoblast cells during early pregnancy. hCG belongs to the glycoprotein hormone (GPH) family and exists as a heterodimer with an alpha and beta subunit. Its beta subunit is unique to hCG, however, its alpha subunit is identical to that of other GPH family members, including luteinizing hormone (LH), follicular stimulating hormone (FSH), and thyroid stimulating hormone (TSH). Due to this similarity to FSH and LH, it can be used as a female fertility treatment, however, hCG can also also stimulate the production of testosterone in the male testes and is sometimes used as a treatment for certain cases of hypogonadism. Unfortunately, this activity has led to hCG abuse by male athletes as a method to increase endogenous testosterone levels despite being listed as a prohibited substance for male athletes by the World Anti-Doping Agency (WADA).

While most anti-doping testing is conducted using mass spectrometric methods, hCG testing is conducted on immunoassay platforms that utilize biotin-streptavidin binding methods (automated analyzers, ELISA). Biotin interference is a well-known confounding factor in biotin-streptavidin immunoassays. Excess biotin in urine or serum binds to streptavidin molecules lowering the sensitivity of the assay. In certain clinical tests that utilize biotin-streptavidin binding, excess biotin can impact immunoassay results in individuals supplementing with biotin at a dose as low as 5 mg/day. Biotin, or vitamin B7, is a coenzyme involved in metabolic processes related to the breakdown of macronutrients. Biotin supplementation is considered safe and non-toxic even at remarkably high doses (<300mg/day) and it is readily available over the counter. Knowing that biotin supplementation is readily available and may be widely used, it is presumable that heavy biotin supplementation may mask illicit hCG use by athletes. To overcome this interference in a clinical setting, a method utilizing streptavidin coated microparticles has been developed to deplete biotin from samples, however this method is costly and not suitable for anti-doping applications.

The goal of this study is to understand whether hCG use can be masked by over-the-counter biotin supplementation, and whether the diafiltration method identified by Sobolevsky and Ahrens is a viable protocol for increased accuracy of hCG testing in urine samples. Additionally, we aim to understand how this potential masking effect is observed in serum samples verses urine samples as biotin is primarily excreted in urine so biotin levels are typically lower in the serum when compared to urine. The study will be conducted in male participants and will include two groups: hCG +oral biotin treatment and hCG + oral placebo treatment. Participants will have seven hCG injections and will be taking an over-the-counter biotin (or placebo) supplement daily from the onset of the study until the final day, 32 days after the first injection.

Experimental Design

Study Drug choriogonadotropin alfa Dose: 250 µg (should equate to between 2000-2300 IU), 2X per week, subcutaneously

Dietary Supplement:

Biotin (20mg), 1x per day, p.o.

Placebo Supplement:

Capsules provided by pharmacy, 1x per day, p.o.

Study Design

Subjects will be divided into two treatment groups:

Cohort 1: hCG treatment, oral biotin supplement Cohort 2: hCG treatment, oral placebo supplement As enrollment occurs, participants will be randomized evenly into one of the two cohorts in 'every other' fashion.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy males aged 18 or older
* Participants must be actively exercising individuals

Exclusion Criteria:

* Individuals below the age of 18 or greater than the age of 55 on the day of enrollment
* Individuals currently enrolled in a registered testing pool for anti-doping purposes
* Individuals unwilling to provide blood or urine samples
* Individuals that are not actively exercising
* Individuals currently using testosterone or undergoing hypogonadism or hypoandrogenism treatment, or have within the previous 3 months
* Individuals at risk for testicular or prostate cancer, as determined by the physician, or with a history of hormone dependent tumors of the reproductive tract and accessory organs (such as prostatic carcinoma, testicular cyst, or breast cancer)
* Individuals that show a high risk of heart attack, blood clots or cardiovascular disease, as defined by the physician, or who are currently using anticoagulant medications
* Individuals with a history of cardiac, renal or hepatic disease, as defined by the physician
* Individuals with a history of prostatic hyperplasia, venous thromboembolism, stroke, edema, or sleep apnea
* Individuals that are diabetic or are currently taking a diabetic medicine
* Individuals with epilepsy
* Individuals with a known allergy to hamster protein or with hypersensitivity to hCG preparations or excipients
* Individuals with a history of aggressive behavior or suicidality

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Identifies as male
Enrollment: 10 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
1. Urinary hCG and biotin concentrations | 6 months
  Urinary hCG concentration will be measured on different analytical platforms (Abbott, Roche, Siemens) that are dependent or not dependent on biotin-streptavidin chemistry for hCG measurement. Urinary biotin concentration will be measured using mass spectrometric techniques. Measured hCG concentrations, especially those during and after the dosing of Ovidrel, will be assessed in combination with the biotin concentration to understand the masking effect of biotin on urinary hCG measurement as it relates to anti-doping.
2. HPT-related hormone measurements in serum; biotin measurements in serum | 6 months
  hCG, LH (luteinizing hormone), FSH (follicle stimulating hormone), testosterone, SHBG (sex hormone binding globulin), and estradiol will be measured in serum before and after treatment with Ovidrel. Changes in each of these compounds will be compared to individual baseline values established prior to Ovidrel use to understand the drug effects. hCG and LH will be measured on analytical platforms known to be affected by biotin interference, and all analytes (including hCG and LH) will be measured on an analytical platform not affected by biotin interference.

SECONDARY OUTCOMES:
1. Detection window of hCG following use | 6 months
  The length of time (following Ovidrel use) that hCG is detectable in urine will be assessed. This will be measured across different analytical platforms and in the presence and absence of biotin supplementation.
2. Urinary testosterone/epitestosterone ratio measurement | 6 months
  The concentrations of testosterone and epitestosterone will be measured using mass spectrometric techniques; results will be compared against measurements obtained at baseline (prior to beginning the Ovidrel dosing).
3. CBC measurements as they relate to the Athlete Biological Passport | 6 months
  Changes from individually established baselines will be assessed for the following complete blood count analytes following Ovidrel dosing: red blood cell count (RBC), hemoglobin concentration (HGB), hematocrit (HCT), mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW), platelet count (PLT), reticulocyte number (RET%), reticulocyte count (RET#), and immature reticulocyte fraction percent (IRF%).

CONTACTS AND LOCATIONS:
Overall Officials: Andre Crouch, MD, Principal Investigator — Sports Medicine Research and Testing Laboratory
Locations (1):
- Sports Medicine Research and Testing Laboratory, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goodrum JM, Nair VS, Moore C, Crouch AK, Eichner D, Miller GD. Impact of Biotin Supplementation on Human Chorionic Gonadotropin Immunoassays Utilizing Biotin-Streptavidin Binding Methods in Urine. Clin Chem. 2023 Jul 5;69(7):754-762. doi: 10.1093/clinchem/hvad060. PMID 37253044